CLINICAL TRIAL: NCT04067882
Title: Prospective Study for the Validation of the Genetic Signature 354849 to Predict the Response to Standard Treatment in Patients With Locally Advanced Cervical Cancer
Brief Title: Validation of the Genetic Signature 354849 as a Prognostic Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trials department, National Institute of Cancerología
Other Study IDs: 019/018/ICI
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cervix Cancer
Keywords: Genetic signature; Treatment response
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples will be collected during the diagnostic biopsy and will be routinely processed by the pathology laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervix cancer: Women older than 18 years with histopathological diagnosis of cervical cancer clinical stage I2-IVA, candidates to receive standard treatment with chemotherapy followed by brachytherapy.
  Interventions: Other: Genetic signature

INTERVENTIONS:
Other: Genetic signature — The RNA will be extracted from the tumor sample with a special kit and a q-PCR will be performed. In order to quantify the genetic expression, the comparative method called Cycle threshold or Crossing point will be used.

SUMMARY:
This prospective study is focused on the validation of the genetic signature of 27 genes as a predictor of the response to concomitant chemotherapy treatment followed by brachytherapy in patients with locally advanced cervical cancer. The genes included are: ZNF238; SAP30; C10orf137; UHRF1; SUZ12; HMGN4; RBBP4; PPP1CB; SLFN11; FLJ39378; ENDOGL1; RECQL; TRPC1; TRIO; DNAH6; GNL3L; SLC36A2; SRP9; RPE; LDOC1L; PUS7L; CCDC89; LOC644921; PLEKHG1; FAM111B; RPRD2 y ETAA16.

DETAILED DESCRIPTION:
There are several studies of genes or genetic signatures associated with the response to treatment in cervical cancer, but so far it has not been possible to standardize the use of any biomarker or biomarker signature as a predictor of the response to treatment with reproducible results. Therefore, there is still a need to develop an effective method to predict the response to chemo-radiotherapy in locally advanced cervical cancer. This prospective study included 189 patients with cervical cancer clinical stages IB2-IVA, without previous treatment.

Tumor samples will be obtained at the confirmatory diagnostic biopsy. All samples will be processed by the pathology laboratory as usual. The RNA will be extracted from the paraffin blocks with the RNeasy FFPE Kit (Qiagen) according to the manufacturer's recommendations. The RNA will be stored at -20°C until use. Quantitative PCR (qPCR) will be performed with the kit High-Capacity cDNA Reverse transcription Kit (Thermo Fisher Scientific). Primers for the 27 genes will be developed. The relative expression will be calculated using the 2- ΔΔCt method, using the expression of β-actin as a normalizing gene.

In order to obtain the prognostic score, the score assigned by the classifier for the sample will be calculated from the 2-ΔΔCt values obtained for each gene. This will be done by a computer-readable medium containing the type expression profiles related to a good and a bad response to the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Cervical Cancer at IB2-IVA FIGO´s clinical stages
* Histology: squamous, adenosquamous or adenocarcinoma
* No previous treatment
* No distance metastases, discard by PET/CT
* Functional State ECOG (Eastern Cooperative Oncology Group) 0-2
* Candidates to receive standard chemoradiotherapy treatment followed by brachytherapy

Exclusion Criteria:

* Previous chemotherapeutic, surgical and/or radiotherapy treatment for female reproductive tract pathologies
* Previous invasive neoplasia (except non-melanoma skin cancer) unless there is complete remission of the disease of 3 years minimum.
* Previous systemic chemotherapy for the current cervical cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the histopathological diagnosis of cervical cancer FIGO's clinical stage IB2-IVA.
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Genetic signature validation | 2 years
  Validate the genetic signature of 27 genes to predict treatment response in patients with cervix cancer.

SECONDARY OUTCOMES:
Predictive values test | 2 years
  Determine sensitivity, specificity and predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: David F Cantú-deLeón, MD, PhD, Principal Investigator — National Cancer Institute of Mexico
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - David Cantu de Leon, Mexico City, Tlalpan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: 2 years
Access Criteria: the data will be shared with scientific and academic institutions or research groups that study the same topic and with the regulatory and ethical authorities that require it, to ensure the quality and accuracy of the data.

REFERENCES:
- [Background] Crosbie EJ, Einstein MH, Franceschi S, Kitchener HC. Human papillomavirus and cervical cancer. Lancet. 2013 Sep 7;382(9895):889-99. doi: 10.1016/S0140-6736(13)60022-7. Epub 2013 Apr 23. PMID 23618600
- [Background] Cohen PA, Jhingran A, Oaknin A, Denny L. Cervical cancer. Lancet. 2019 Jan 12;393(10167):169-182. doi: 10.1016/S0140-6736(18)32470-X. PMID 30638582
- [Background] Bhatla N, Aoki D, Sharma DN, Sankaranarayanan R. Cancer of the cervix uteri. Int J Gynaecol Obstet. 2018 Oct;143 Suppl 2:22-36. doi: 10.1002/ijgo.12611. PMID 30306584
- [Background] Todo Y, Watari H. Concurrent chemoradiotherapy for cervical cancer: background including evidence-based data, pitfalls of the data, limitation of treatment in certain groups. Chin J Cancer Res. 2016 Apr;28(2):221-7. doi: 10.21147/j.issn.1000-9604.2016.02.10. PMID 27199520
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Leath CA 3rd, Monk BJ. Twenty-first century cervical cancer management: A historical perspective of the gynecologic oncology group/NRG oncology over the past twenty years. Gynecol Oncol. 2018 Sep;150(3):391-397. doi: 10.1016/j.ygyno.2018.06.023. Epub 2018 Jun 27. PMID 29954593
- [Background] Thomas GM. Improved treatment for cervical cancer--concurrent chemotherapy and radiotherapy. N Engl J Med. 1999 Apr 15;340(15):1198-200. doi: 10.1056/NEJM199904153401509. No abstract available. PMID 10202172
- [Background] Lakosi F, de Cuypere M, Viet Nguyen P, Jansen N, Warlimont B, Gulyban A, Gennigens C, Seidel L, Delbecque K, Coucke P, Hermesse J, Kridelka F. Clinical efficacy and toxicity of radio-chemotherapy and magnetic resonance imaging-guided brachytherapy for locally advanced cervical cancer patients: A mono-institutional experience. Acta Oncol. 2015;54(9):1558-66. doi: 10.3109/0284186X.2015.1062542. Epub 2015 Sep 25. PMID 26406152
- [Background] Chuang L, Kanis MJ, Miller B, Wright J, Small W Jr, Creasman W. Treating Locally Advanced Cervical Cancer With Concurrent Chemoradiation Without Brachytherapy in Low-resource Countries. Am J Clin Oncol. 2016 Feb;39(1):92-7. doi: 10.1097/COC.0000000000000222. PMID 26398064
- [Background] Chemoradiotherapy for Cervical Cancer Meta-analysis Collaboration (CCCMAC). Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: individual patient data meta-analysis. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD008285. doi: 10.1002/14651858.CD008285. PMID 20091664
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Marita A, Ordeanu C, Rancea A, Nicolae T, Nagy VM. Long-term survival following neoadjuvant chemotherapy and concomitant radiochemotherapy in locally advanced cervical cancer: results of the Oncology Institute "Prof. Dr. Ion Chiricuta" experience. J Med Life. 2018 Jan-Mar;11(1):42-50. PMID 29696064
- [Background] Yin KC, Lu CH, Lin JC, Hsu CY, Wang L. Treatment outcomes of locally advanced cervical cancer by histopathological types in a single institution: A propensity score matching study. J Formos Med Assoc. 2018 Oct;117(10):922-931. doi: 10.1016/j.jfma.2018.07.002. Epub 2018 Jul 17. PMID 30025761
- [Background] Horikawa N, Baba T, Matsumura N, Murakami R, Abiko K, Hamanishi J, Yamaguchi K, Koshiyama M, Yoshioka Y, Konishi I. Genomic profile predicts the efficacy of neoadjuvant chemotherapy for cervical cancer patients. BMC Cancer. 2015 Oct 19;15:739. doi: 10.1186/s12885-015-1703-1. PMID 26482555
- [Background] Moreno-Acosta P, Carrillo S, Gamboa O, Romero-Rojas A, Acosta J, Molano M, Balart-Serra J, Cotes M, Rancoule C, Magne N. Novel predictive biomarkers for cervical cancer prognosis. Mol Clin Oncol. 2016 Dec;5(6):792-796. doi: 10.3892/mco.2016.1055. Epub 2016 Oct 19. PMID 28101358
- [Background] Chen Q, Tian WJ, Huang ML, Liu CH, Yao TT, Guan MM. Association Between HIF-1 Alpha Gene Polymorphisms and Response in Patients Undergoing Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer. Med Sci Monit. 2016 Sep 5;22:3140-6. doi: 10.12659/msm.897486. PMID 27593081
- [Background] Fernandez-Retana J, Lasa-Gonsebatt F, Lopez-Urrutia E, Coronel-Martinez J, Cantu De Leon D, Jacobo-Herrera N, Peralta-Zaragoza O, Perez-Montiel D, Reynoso-Noveron N, Vazquez-Romo R, Perez-Plasencia C. Transcript profiling distinguishes complete treatment responders with locally advanced cervical cancer. Transl Oncol. 2015 Apr;8(2):77-84. doi: 10.1016/j.tranon.2015.01.003. PMID 25926073
- [Background] Zwenger AO, Grosman G, Iturbe J, Leone J, Vallejo CT, Leone JP, Verdera PP, Perez JE, Leone BA. Expression of ERCC1 and TUBB3 in locally advanced cervical squamous cell cancer and its correlation with different therapeutic regimens. Int J Biol Markers. 2015 Jul 22;30(3):e301-14. doi: 10.5301/jbm.5000161. PMID 26165688
- [Background] Wen YF, Cheng TT, Chen XL, Huang WJ, Peng HH, Zhou TC, Lin XD, Zeng LS. Elevated circulating tumor cells and squamous cell carcinoma antigen levels predict poor survival for patients with locally advanced cervical cancer treated with radiotherapy. PLoS One. 2018 Oct 10;13(10):e0204334. doi: 10.1371/journal.pone.0204334. eCollection 2018. PMID 30303986
- See also: Ferlay J, Ervik M, Lam F, Colombet M, Mery L, Piñeros M, Znaor A, Soerjomataram I, B.F. Global Cancer Observatory: Cancer Today — https://gco.iarc.fr/today/home
- See also: World Health Organitation. Human papillomavirus (HPV) and cervical cancer. — http://www.who.int/news-room/fact-sheets/detail/human-papillomavirus-(hpv)-and-cervical-cancer